CLINICAL TRIAL: NCT03810040
Title: Effect of Degranulation Needle on the Rate Good Embryo in IVF
Brief Title: Effect of Degranulation Needle With Different Diameters on the Rate Good Embryo in IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123456
Record Dates: First submitted 2018-07-05; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Embryo
Keywords: Embryos quality; In vitro fertilization; Denuding pipette

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Odd-numbered days (Active Comparator): Once odd-numbered days the zytoges of IVF cycle were collected. The 140 microns denuding pipette was used.
  Interventions: Device: 140 microns denuding pipette
- Even-numbered days (Experimental): Once even-numbered days the zytoges of IVF cycle were collected. The 150 microns denuding pipette was used.
  Interventions: Device: 150 microns denuding pipette

INTERVENTIONS:
Device: 140 microns denuding pipette — the degranulated needle size was 140 microns
  Arms: Odd-numbered days
Device: 150 microns denuding pipette — the degranulated needle size was 150 microns
  Arms: Even-numbered days

SUMMARY:
Good-quality embryos are critical for the success of in vitro fertilization (IVF). But, to date, there is no report of the effect of different diameters denuding pipette on the embryos quality. To investigate the effect of denuding pipette in IVF outcomes, we plan to recruit women undergoing IVF treatment cycles and classified them into two groups according to the different diameters. Consequently, the rate of fertilization, zygotes cleaved, top quality embryos on D3, and blastocysts obtained were recorded.

DETAILED DESCRIPTION:
Good-quality embryos are critical for the success of in vitro fertilization (IVF). But, to date, there is no report of the effect of different diameters denuding pipette on the embryos quality. To investigate the effect of denuding pipette in IVF outcomes, we plan to recruit women undergoing IVF treatment cycles and classified them into two groups according to the different diameters. The participants were divided into two group. Odd-numbered days the zygotes were degranulated with the 140 microns needles. Even-numbered days the zygotes were degranulated with the 150 microns needles. Consequently, the rate of fertilization, zygotes cleaved, top quality embryos on D3, and blastocysts obtained were recorded.

ELIGIBILITY:
Inclusion Criteria:

* first cyele of IVF treatment

Exclusion Criteria:

* oocyte number less than 4
* oocyte number over than 25

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
quality of embryo | one year
  embryo quality assessed by good embryo rate

SECONDARY OUTCOMES:
clinical outcome - clinical prengancy rate | three years
  clinical prengancy rate

CONTACTS AND LOCATIONS:
Overall Officials: jin ni, Study Director — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No